CLINICAL TRIAL: NCT03786614
Title: Antidepressant Discontinuation in Treatment Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rifaat S. El-Mallakh, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.1351
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Treatment Resistant Depression
Keywords: treatment resistant depression; serotonergic antidepressants; short form of serotonin transporter
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person performing the data collection (rater) will be blind to the randomization of the patient for the entire duration of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation arm (Active Comparator): This group will be discontinued from serotonergic antidepressants and shifting them to other categories of antidepressants, i.e., medications that work through dopamine or nor-epinephrine, or by reducing the serotonin signal rather than increasing synaptic serotonin, as might be accomplished with low dose, sub-anti-psychotic doses of some second-generation anti-psychotics.
  Interventions: Other: Discontinuation of serotonergic antidepressants
- Continuation arm (Active Comparator): This group will continue taking serotonergic antidepressants which is the standard care of treatment.
  Interventions: Other: Continuation of serotonergic medications

INTERVENTIONS:
Other: Discontinuation of serotonergic antidepressants — Discontinuation of serotonergic antidepressants and possibly shift to other antidepressant categories that were proven to be effective in treating depression such as pramipexole, bupropion, quetiapine, lurasidone, brexpipazole. Additionally, subjects will have access to other treatment measures of treating treatment resistant depression.
  Arms: Discontinuation arm
Other: Continuation of serotonergic medications — Continuation of serotonergic medications which is the standard care of treatment. Additionally, subjects will have access to other treatment measures of treating treatment resistant depression.
  Arms: Continuation arm

SUMMARY:
The purpose of this study is to compare the effects on depressive symptoms of subjects who discontinue serotonergic antidepressants (a certain type of antidepressant, such as Prozac, that works on serotonin receptors in the brain) with the effects on depressive symptoms of subjects who continue to take serotonergic antidepressants. During this study, subjects will also be presented with the opportunity to undergo genetic testing for the serotonin gene transporter which has a short or long form. This is being done because it has been demonstrated that genetic testing improves outcome while treating treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be a man or woman 18 to 70 years of age, inclusive.
* Subject must meet criteria for a major depressive disorder as confirmed by the Mini International Neuropsychiatric Interview [MINI].
* Subjects must have a current Treatment-Resistant Depression as defined below.
* Subjects must have been taking serotonergic antidepressants (serotonin reuptake inhibitor or monoamine oxidase inhibitor) for at least 2 years but not more than 4 years, and have failed 2 previous medication trial for the current episode. Current Montgomery-Åsberg Depression Rating Scale [MADRS] score must be equal to or more than 25.
* Subject must be medically stable.
* Female subjects must have a negative urine pregnancy test at screening, and agree to avoid pregnancy during the study.
* Each subject must sign an informed consent form indicating that he/she understands the purpose of the study and the procedures required and are willing to participate in the study.
* Subject must be able to participate in symptom measurement.

Exclusion Criteria:

* Subject has a current Diagnostic and Statistical Manual of Mental Disorders-5 [DSM-5] diagnosis of bipolar disorder or has a positive screening for bipolar disorder by Mini International Neuropsychiatric Interview [MINI] or Mood Disorder Questionnaire [MDQ].
* Subject has a current DSM-5 diagnosis of schizophrenia, schizoaffective disorder, autistic disorder, or intellectual disability.
* Subject has a substance use disorder (except for nicotine or cannabis) within 3 months prior to screening or has a positive drug screen test for any recreational drugs at the time of screening with the exception of Cannabis.
* Subject has evidence of any clinically significant, unstable medical problems that may create a safety risk for a subject, interfere with study participation, or make results difficult to interpret.
* Subject is at imminent risk of suicide according to the investigator's clinical judgment and/or a Columbia-Suicide Severity Rating Scale (C-SSRS) 3 or more at any time in the study.
* Subject is a woman who is pregnant, breast-feeding or planning to become pregnant while enrolled in the study.
* Subject has any condition (according to the investigator) for which participation will not be the best interest for the subject or it can prevent, limit or confound the protocol-specified assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the difference of response as measured by the Montgomery-Åsberg Depression Rating Scale [MADRS] between both arms. | From baseline and every visit [every 4 weeks] to the end of the study. [6 months]
  The MADRS is a psychiatric scale to assess the depressive symptoms from the patient's prospective. The final score ranges from 0 to 60 with 0 indicating no depression and higher scores indicating greater depression. The final scores will be evaluated with a non-paired, two-tailed t-test.
Comparing the difference of response as measured by the Montgomery-Åsberg Depression Rating Scale [MADRS] between subjects with low expressing alleles and high expressing alleles of the serotonin gene transporter. | End of study [6 months].
  Genetic testing for the serotonin transporter gene will be done for every patient in the study. All subjects with homozygous and heterozygous low expression alleles will be combined as one group, and all high expression subjects will be the other group. One-way ANOVAs will be conducted for each genotype group, with genotype group as the independent variable (IV) and MADRS scores as the dependent variables (DV).

SECONDARY OUTCOMES:
Evaluating changes in levels of anxiety as measured by the Hamilton Anxiety Rating Scale [HAM-A] between both arms. | From baseline and every visit [every 4 weeks] to the end of the study. [6 months]
  The HAM-A will be collected to assess changes in anxiety levels from the patient's prospective. It ranges from 0 to 56 with greater scores indicating more anxiety. The final scores will be evaluated with a non-paired, two-tailed t-test.
Evaluating the difference of response as measured by the Columbia Suicide Severity Rating Scale [C-SSRS] between both arms. | From baseline and every visit [every 4 weeks] to the end of the study. [6 months]
  The C-SSRS is a psychiatric scale to assess suicidality. It ranges from 0 to 5 with 0 indicating no suicidal ideas and higher scores indicating greater suicidal ideas. The final scores will be evaluated with a non-paired, two-tailed t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Rifaat S. El-Mallakh, MD, Principal Investigator — University of Louisville, Department of Psychiatry and Behavioral Sciences
Locations (1):
- University of Louisville, Department of Psychiatry and Behavioral Sciences, Louisville, Kentucky, United States